CLINICAL TRIAL: NCT04821531
Title: Impact of Adding a Self-guided Exercise Program on Functional Outcomes Among Hospitalized COVID-19 Patients: A Randomized Prospective Study
Brief Title: Feasibility of a Self-guided Exercise Program Among Hospitalized COVID-19 Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID patients admitted to the hospital during the study dates did NOT have the criteria to enter the study(i.e they were too medically unstable) or their hospital stay was too short to conduct a before and after assessment
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-12575
Record Dates: First submitted 2021-03-11; First posted 2021-03-29 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Corona Virus Infection
Keywords: coronavirus; covid; covid-19; covid19; corona
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blind(outcome assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PT Pal (Experimental): Experimental Arm-PT PAL Participants randomized into this arm will receive exercise instructions via Pt_PAL. PT PAL is a mobile health technology used to facilitate communications between Care teams and patients, by allowing the team to send web-based exercise routines, surveys and educational materials. The PT Pal app captures patient activity adherence and reports
  Interventions: Other: PT Pal
- Exercise Manual (Active Comparator): Control Arm- Exercise Manual Participants randomized into this arm will use the exercise manual to obtain their exercise instructions
  Interventions: Other: Exercise Manual

INTERVENTIONS:
Other: PT Pal — Patients will be guided through individualized exercises that will be selected by their primary physical therapists. The exercises aim to improve lung function, maintain joint flexibility, muscle strength balance and mobility
  Arms: PT Pal
Other: Exercise Manual — Patients will be guided through individualized exercises that will be selected by their primary physical therapists. The exercises aim to improve lung function, maintain joint flexibility, muscle strength, balance and mobility
  Arms: Exercise Manual

SUMMARY:
The investigators' aim is to conduct a study looking into safety and feasibility study of Covid patients participating in a self-guided exercises program while admitted to the hospital. The investigators will test 2 forms of exercise instruction, one using an exercise phone-based application, and the other a printed exercise manual.

DETAILED DESCRIPTION:
The COVID-19 pandemic has resulted in significant morbidity and mortality throughout the world. As of March 16, 2021 there were over 119 million confirmed COVID-19 cases and 2.6 million deaths globally. The majority of COVID-19 cases are mild to moderate, resulting in symptom resolution within 6 weeks of symptom onset.

Following moderate to severe COVID-19 infections, functional impairments are likely to be dominated by peripheral muscle dysfunction (due to deconditioning and decreased lean body mass, ICU neuropathy, fatigue and the effects of hypoxemia), respiratory muscle dysfunction (dysfunctional breathing pattern, DBP, and exercise-induced laryngeal obstruction), cardiac impairment and deconditioning, and psychosocial factors (anxiety, depression, guilt, sleep disturbance and dependency).

Physical exercise has proven to be an effective therapy for most chronic diseases and microbial infections with preventive or therapeutic benefits involving the primary immunological mediators and/or anti-inflammatory properties. Another mechanism is that it can counteract the effect of prolonged bedrest by preventing the decline in muscle strength, muscle mass loss , reduce exaggerated cardiac response to exercise, reduce thromboembolism, and improve lung function. Prior research in COPD patients have shown that early pulmonary rehabilitation showed reductions in mortality, length of stay and readmission.

There has been some concern among physicians about allowing patients with COVID-19 to exercise. This is also of concern to all practitioners of Rehabilitation Medicine and the investigators seek to understand the risks better. This research group is currently concluding another retrospective study of 988 COVID-19 patients that suggest that not only is exercise safe, but increasing the number of exercise interventions improves the functional status of the patients and may reduce mortality.

As the next step, the investigators propose a 12-month, single blind feasibility study to determine if adding a self-guided exercise to a patient population already receiving two 30-minutes/week therapy can improve the patient's overall functional and cognitive outcomes. The overall hypothesis is that COVID-19 patients admitted to the hospital with mild to moderate disease can safely perform these exercises and improve their physical and cognitive functioning. The objective in performing this study is to examine feasibility as well as obtain preliminary data to design future RCT studies in this or other similar diseases. The self-guided exercise program was developed by the Department of Rehabilitation at Montefiore during the initial COVID-19 surge. The manual has been published in the Journal for the International Society of Physical and Rehabilitation Medicine and has been distributed through many medical society websites. COVID-19 patients admitted to the Montefiore Hospital have been receiving the exercise manual upon discharge for the past 9 months. The exercises in the program are divided into 3 levels. The initial level focuses on prevention of lung complication associated with COVID-19, and prevention of contracture in the large joints associated with bedrest. The next level focuses on improving sitting tolerance, strengthening limb and accessory muscles of breathing. The final level works on standing balance, large muscle strengthening, and building cardiopulmonary endurance The investigators will test 2 modes of delivery, one using the printed exercise manual and the other using Pt PAL, a mobile health technology application. Pt PAL can facilitate communication between the care team and patients, and allows the team to send from their web-portal, exercise routines, surveys and educational material to the patient's mobile device. The Pt PAL app then captures the patient activity adherence, and reports those results back to the team including a graphical summary about patients' condition and activity. The investigators have successfully applied Pt PAL exercise program to other patient populations (e.g., heart failure patients) in Montefiore Medical Center, and the app has received regulatory approval at Montefiore.

The research team composed of Rehabilitation Medicine physician, Internal Medicine specialist, rehabilitation therapists, nursing, medical students and research staff are very well positioned to carry out a study of this nature effectively and safely to its conclusion.

The investigators will assess the changes in the following measures

1. Activity Measure for Post-Acute Care (AM-PAC)12 which was developed to examine basic mobility and daily activity functional activities important to adults.
2. St George's Respiratory function questionnaire to assess pulmonary function. It is scored for symptoms, physical activity, and impact domains
3. Short Physical Performance Battery (SPPB ) is a series of physical performance tests used in older persons to assess lower extremity function, balance and mobility and is predictive of a broad range of adverse outcomes, including mortality, incident disability, falls, hospitalization and healthcare utilization.
4. The Picture Memory Impairment Screen is a brief, 4-item free and cued recall test of memory that uses pictures to overcome many of the educational, cultural, and logistical barriers to cognitive screening in clinical settings and is nondiscriminatory with regard to culture and literacy.
5. The Paper Match Stimuli, a rapid paper test that can be administered under 3 minutes correlate predominantly with brain regions mediating information processing speed (i.e., basal ganglia) and executive functions (i.e., dorsolateral prefrontal and parietal cortex
6. The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression, which can help identify patients whose motivation for exercise may be impacted by depression

ELIGIBILITY:
Inclusion

* COVID-19 Positive by PCR testing
* Adults aged 50-75
* Patients evaluated by Rehabilitation team and found appropriate for the study
* Able to read and understand English or Spanish
* Have access to a smartphone

Exclusion

* Pregnant patients
* Patients with dementia or cognitive dysfunction
* Patients who exhibit poor safety or unsafe behavior
* Patients who need high flow oxygen, rebreather or any form of ventilatory support
* Patients with chest tubes or similar attachments

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-02-23 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Adherence: Number of Days patient exercises independently at least 1 time a day | 1 year
Recruitment , Implementation and Retention: number of patients contacted, enrolled and completed study | 1 year
Safety: Number of adverse health events | 1 year

SECONDARY OUTCOMES:
Activity Measure for Post-Acute Care (AM-PAC). | 1 year
  The range is 6-24; higher scores reflect better mobility
St George's Respiratory function questionnaire | 1 year
  The range is 0 to 100; higher scores worse.
Short Physical Performance Battery (SPPB ) | 1 year
  The scores range from 0-12, higher scores reflect better lower extremity function.
The Picture Memory Impairment Screen | 1 year
  The scores range from 0-8, higher scores reflect better memory function.
The Paper Match Stimuli. | 1 year
  The scores range from 0-52, higher scores better processing speed and executive function.
The Beck Depression Inventory (BDI). | 1 year
  The scores range from 0-63. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depression.
Discharge Destination | 1 year
  Percentage of patients being discharged home, versus those who require discharge to rehabilitation hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Anne Felice Ambrose, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No